CLINICAL TRIAL: NCT03447002
Title: Urine Levels of Metanephrin and Normetanephrin in Patients With Frequent Ventricular Premature Complex
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Burak Cesur, burak cesur, TC Erciyes University
Other Study IDs: ErciyesU
Record Dates: First submitted 2018-02-19; First posted 2018-02-27 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Premature Ventricular Contraction
Keywords: premature; pvc
MeSH Terms: conditions — Ventricular Premature Complexes; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 24 hours urine levels metanephrine and normetanephrine — 24 hours rhythm recording and 24 hours urine measurement
  Other Names: rhythm recording

SUMMARY:
Enhanced automaticity process is the underlying mechanism for arrhythmias due to excess catecholamines. Catecholamines may increase in patients with PVC. Metabolites of catecholamines are metanephrine and normetanephrine. Our aim is to measure 24 hours urine levels of metanephrine and normetanephrine.

DETAILED DESCRIPTION:
Premature ventricular complex is a very frequent arrhythmia. Suggested mechanisms for PVCs are reentry, triggered activity, and enhanced automaticity. Enhanced automaticity process is the underlying mechanism for arrhythmias due to excess catecholamines. Catecholamines may increase in patients with PVC. Half-lives of catecholamines are very short and rather changeable. Therefore, 24 hours urine levels of catecholamines are the more sensitive than plasma levels. Metabolites of catecholamines are metanephrine and normetanephrine. Our aim is to measure 24 hours urine levels of metanephrine and normetanephrine.

ELIGIBILITY:
Inclusion Criteria:

* PVC's rate is more than % 5 in 24 hours rhythm recording

Exclusion Criteria:

* ischemic heart disease
* hyperthyroidism
* patients with low ejection fraction

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with % 5 or higher frequents premature ventricular complex in 24 hours rhythm recording will be taken our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
metanephrine and normetanephrine levels | about 10 months
  metanephrine and normetanephrine levels asociated premature ventricular complex frequents

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes university Yilmaz- mehmet öztaşkın heart hospital, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Im SI, Park KM, Park SJ, Kim JS, On YK. New electrocardiographic criteria for predicting successful ablation of premature ventricular contractions from the right coronary cusp. Int J Cardiol. 2016 Dec 1;224:199-205. doi: 10.1016/j.ijcard.2016.09.029. Epub 2016 Sep 16. PMID 27657474
- [Background] Bradfield JS, Homsi M, Shivkumar K, Miller JM. Coupling interval variability differentiates ventricular ectopic complexes arising in the aortic sinus of valsalva and great cardiac vein from other sources: mechanistic and arrhythmic risk implications. J Am Coll Cardiol. 2014 May 27;63(20):2151-2158. doi: 10.1016/j.jacc.2014.02.551. Epub 2014 Mar 19. PMID 24657687
- [Derived] Cesur B, Elcik D, Cetinkaya Z, Kelesoglu S, Karabiyik U, Inanc MT, Kalay N, Ergin A, Topsakal R. Association between excess catecholamine synthesis and polymorphic premature ventricular contraction. J Electrocardiol. 2024 Jan-Feb;82:59-63. doi: 10.1016/j.jelectrocard.2023.11.010. Epub 2023 Nov 26. PMID 38035655